CLINICAL TRIAL: NCT06979986
Title: Systematically Mediastinal Lymph Node Dissection (SLND) Versus Non-Dissection Following Endoscopic Submucosal Dissection (ESD) for T1a Stage Esophageal Squamous Cell Carcinoma
Brief Title: SLND Versus Non-Dissection Following ESD for T1a Stage Esophageal Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FJCHTOSP-1
Record Dates: First submitted 2025-05-01; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic Submucosal Dissection with Systematically mediastinal Lymph Node Dissection (Experimental): T1a Stage Esophageal Squamous Cell Carcinoma undergo Endoscopic Submucosal Dissection with Systematically mediastinal Lymph Node Dissection
  Interventions: Procedure: Endoscopic Submucosal Dissection with Systematically mediastinal Lymph Node Dissection
- Endoscopic Submucosal Dissection without Systematically mediastinal Lymph Node Dissection (Placebo Comparator): T1a Stage Esophageal Squamous Cell Carcinoma just recieve Endoscopic Submucosal Dissection treatment, not undergo Systematically mediastinal Lymph Node Dissection
  Interventions: Procedure: Endoscopic Submucosal Dissection without SLND

INTERVENTIONS:
Procedure: Endoscopic Submucosal Dissection with Systematically mediastinal Lymph Node Dissection — Participants will be evaluated for inclusion criteria and exclusion criteria, and then sign informal consent if desired. Participants will be randomly assigned to the intervention according to a prepared random tables. Participants in the SLND group will receive Endoscopic Submucosal Dissection with systematically mediastinal lymph node dissection
  Arms: Endoscopic Submucosal Dissection with Systematically mediastinal Lymph Node Dissection
Procedure: Endoscopic Submucosal Dissection without SLND — Participants will be evaluated for inclusion criteria and exclusion criteria, and then sign informal consent if desired. Participants will be randomly assigned to the intervention according to a prepare random tables. Participants in the non-SLND group will just receive Endoscopic Submucosal Dissection treatment, not undergo Systematically mediastinal Lymph Node Dissection.
  Arms: Endoscopic Submucosal Dissection without Systematically mediastinal Lymph Node Dissection

SUMMARY:
This is a study from Fujian Cancer Hospital Thoracic of Surgery Project, numbered as FJCHTOSP-1. Systematically mediastinal Lymph Node Dissection (SLD) Versus Non-Dissection Following Endoscopic Submucosal Dissection (ESD) for T1a Stage Esophageal Squamous Cell Carcinoma: a single-center, prospective clinical trial.

DETAILED DESCRIPTION:
Participants will be evaluated for inclusion criteria and exclusion criteria, and then sign informal consent if desired. Participants will be randomly assigned to the intervention according to a prepared random tables. Participants in the systematically mediastinal lymph node dissection (SLND) group will receive systematically mediastinal lymph node dissection, while those in the non-SLND group will not receive mediastinal lymph node dissection. The primary endpoint is 3-year disease-free survival (DFS).

The sample size are estimated with reference to investigators' previous data, in which the 3-year DFS was 62.7% for patients diagnosed with T1a Stage Esophageal Squamous Cell Carcinoma and underwent Endoscopic Submucosal Dissection without SLND. Investigators assumed that if 3-year DFS of patients in SLND group was over 80%, then investigatorswould deem the SLND group to be superior to the non-SLND group. The sample size are estimated to be 102. Therefore, the total number of patients enrolled are designed to be 102.

ELIGIBILITY:
Inclusion Criteria:

* Clinical stage T1aN0M0.
* A lesion detected on Endoscopic Ultrasound featured as T1a stage.
* Age 18 to 75.
* Patients who have signed the informed consent form.

Exclusion Criteria:

* • Other than invasive adenocarcinoma by pathological analysis.

  * Not complete resected or curative intent.
  * Patients who have history of other malignant tumors.
  * Patients who have history of thoracic surgery.
  * Patients who have received radiation, chemotherapy or other treatments previously.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
DFS | From enrollment to the end of treatment at 3 years
  disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Weimin Fang, Principal Investigator

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared due to privacy regulations and restrictions stipulated by the ethics committee approval. Research participants were not informed during the consent process that their data might be widely shared. Additionally, this trial involves sensitive medical information that carries potential re-identification risks even after de-identification procedures. However, researchers interested in specific analyses are welcome to discuss potential collaboration through appropriate data use agreements.

REFERENCES:
- [Result] Nishihira T, Hirayama K, Mori S. A prospective randomized trial of extended cervical and superior mediastinal lymphadenectomy for carcinoma of the thoracic esophagus. Am J Surg. 1998 Jan;175(1):47-51. doi: 10.1016/s0002-9610(97)00227-4. PMID 9445239
- [Result] Altorki N, Kent M, Ferrara C, Port J. Three-field lymph node dissection for squamous cell and adenocarcinoma of the esophagus. Ann Surg. 2002 Aug;236(2):177-83. doi: 10.1097/00000658-200208000-00005. PMID 12170022
- [Result] Tong DK, Law S, Kwong DL, Chan KW, Lam AK, Wong KH. Histological regression of squamous esophageal carcinoma assessed by percentage of residual viable cells after neoadjuvant chemoradiation is an important prognostic factor. Ann Surg Oncol. 2010 Aug;17(8):2184-92. doi: 10.1245/s10434-010-0995-2. Epub 2010 Mar 9. PMID 20217248
- [Result] Tachibana M, Kinugasa S, Yoshimura H, Dhar DK, Nagasue N. Extended esophagectomy with 3-field lymph node dissection for esophageal cancer. Arch Surg. 2003 Dec;138(12):1383-9; discussion 1390. doi: 10.1001/archsurg.138.12.1383. PMID 14662544
- [Result] Ando N, Ozawa S, Kitagawa Y, Shinozawa Y, Kitajima M. Improvement in the results of surgical treatment of advanced squamous esophageal carcinoma during 15 consecutive years. Ann Surg. 2000 Aug;232(2):225-32. doi: 10.1097/00000658-200008000-00013. PMID 10903602
- [Result] Hsu PK, Huang CS, Wang BY, Wu YC, Hsu WH. Survival benefits of postoperative chemoradiation for lymph node-positive esophageal squamous cell carcinoma. Ann Thorac Surg. 2014 May;97(5):1734-41. doi: 10.1016/j.athoracsur.2013.12.041. Epub 2014 Mar 6. PMID 24612702
- [Result] Hsu PK, Wang BY, Huang CS, Wu YC, Hsu WH. Prognostic factors for post-recurrence survival in esophageal squamous cell carcinoma patients with recurrence after resection. J Gastrointest Surg. 2011 Apr;15(4):558-65. doi: 10.1007/s11605-011-1458-1. Epub 2011 Feb 15. PMID 21327531
- [Result] Merkow RP, Bilimoria KY, Keswani RN, Chung J, Sherman KL, Knab LM, Posner MC, Bentrem DJ. Treatment trends, risk of lymph node metastasis, and outcomes for localized esophageal cancer. J Natl Cancer Inst. 2014 Jul 16;106(7):dju133. doi: 10.1093/jnci/dju133. Print 2014 Jul. PMID 25031273
- [Result] Chen J, Wu S, Zheng X, Pan J, Zhu K, Chen Y, Li J, Liao L, Lin Y, Liao Z. Cervical lymph node metastasis classified as regional nodal staging in thoracic esophageal squamous cell carcinoma after radical esophagectomy and three-field lymph node dissection. BMC Surg. 2014 Dec 19;14:110. doi: 10.1186/1471-2482-14-110. PMID 25527100
- [Result] Li H, Yang S, Zhang Y, Xiang J, Chen H. Thoracic recurrent laryngeal lymph node metastases predict cervical node metastases and benefit from three-field dissection in selected patients with thoracic esophageal squamous cell carcinoma. J Surg Oncol. 2012 May;105(6):548-52. doi: 10.1002/jso.22148. Epub 2011 Nov 21. PMID 22105736
- [Result] Tachibana M, Kinugasa S, Yoshimura H, Shibakita M, Tonomoto Y, Dhar DK, Nagasue N. Clinical outcomes of extended esophagectomy with three-field lymph node dissection for esophageal squamous cell carcinoma. Am J Surg. 2005 Jan;189(1):98-109. doi: 10.1016/j.amjsurg.2004.10.001. PMID 15701501
- [Result] Tabira Y, Kitamura N, Yoshioka M, Tanaka M, Nakano K, Toyota N, Mori T. Significance of three-field lymphadenectomy for carcinoma of the thoracic esophagus based on depth of tumor infiltration, lymph nodal involvement and survival rate. J Cardiovasc Surg (Torino). 1999 Oct;40(5):737-40. PMID 10597014
- [Result] Ma GW, Situ DR, Ma QL, Long H, Zhang LJ, Lin P, Rong TH. Three-field vs two-field lymph node dissection for esophageal cancer: a meta-analysis. World J Gastroenterol. 2014 Dec 21;20(47):18022-30. doi: 10.3748/wjg.v20.i47.18022. PMID 25548502
- [Result] Ye K, Xu JH, Sun YF, Lin JA, Zheng ZG. Characteristics and clinical significance of lymph node metastases near the recurrent laryngeal nerve from thoracic esophageal carcinoma. Genet Mol Res. 2014 Aug 25;13(3):6411-9. doi: 10.4238/2014.August.25.4. PMID 25158259
- [Result] Sgourakis G, Gockel I, Lang H. Endoscopic and surgical resection of T1a/T1b esophageal neoplasms: a systematic review. World J Gastroenterol. 2013 Mar 7;19(9):1424-37. doi: 10.3748/wjg.v19.i9.1424. PMID 23539431
- [Result] Fujita H, Sueyoshi S, Yamana H, Shinozaki K, Toh U, Tanaka Y, Mine T, Kubota M, Shirouzu K, Toyonaga A, Harada H, Ban S, Watanabe M, Toda Y, Tabuchi E, Hayabuchi N, Inutsuka H. Optimum treatment strategy for superficial esophageal cancer: endoscopic mucosal resection versus radical esophagectomy. World J Surg. 2001 Apr;25(4):424-31. doi: 10.1007/s002680020053. PMID 11344392
- [Result] Katada C, Muto M, Momma K, Arima M, Tajiri H, Kanamaru C, Ooyanagi H, Endo H, Michida T, Hasuike N, Oda I, Fujii T, Saito D. Clinical outcome after endoscopic mucosal resection for esophageal squamous cell carcinoma invading the muscularis mucosae--a multicenter retrospective cohort study. Endoscopy. 2007 Sep;39(9):779-83. doi: 10.1055/s-2007-966761. PMID 17703385
- [Result] Moriya H, Ohbu M, Kobayashi N, Tanabe S, Katada N, Futawatari N, Sakuramoto S, Kikuchi S, Okayasu I, Watanabe M. Lymphatic tumor emboli detected by D2-40 immunostaining can more accurately predict lymph-node metastasis. World J Surg. 2011 Sep;35(9):2031-7. doi: 10.1007/s00268-011-1143-2. PMID 21667194
- [Result] Yamashina T, Ishihara R, Nagai K, Matsuura N, Matsui F, Ito T, Fujii M, Yamamoto S, Hanaoka N, Takeuchi Y, Higashino K, Uedo N, Iishi H. Long-term outcome and metastatic risk after endoscopic resection of superficial esophageal squamous cell carcinoma. Am J Gastroenterol. 2013 Apr;108(4):544-51. doi: 10.1038/ajg.2013.8. Epub 2013 Feb 12. PMID 23399555
- [Result] Tachibana M, Hirahara N, Kinugasa S, Yoshimura H. Clinicopathologic features of superficial esophageal cancer: results of consecutive 100 patients. Ann Surg Oncol. 2008 Jan;15(1):104-16. doi: 10.1245/s10434-007-9604-4. Epub 2007 Sep 22. PMID 17891442
- [Result] Choi JY, Park YS, Jung HY, Ahn JY, Kim MY, Lee JH, Choi KS, Kim DH, Choi KD, Song HJ, Lee GH, Cho KJ, Kim JH. Feasibility of endoscopic resection in superficial esophageal squamous carcinoma. Gastrointest Endosc. 2011 May;73(5):881-9, 889.e1-2. doi: 10.1016/j.gie.2010.12.028. Epub 2011 Mar 9. PMID 21392755
- [Result] Eguchi T, Nakanishi Y, Shimoda T, Iwasaki M, Igaki H, Tachimori Y, Kato H, Yamaguchi H, Saito D, Umemura S. Histopathological criteria for additional treatment after endoscopic mucosal resection for esophageal cancer: analysis of 464 surgically resected cases. Mod Pathol. 2006 Mar;19(3):475-80. doi: 10.1038/modpathol.3800557. PMID 16444191
- [Result] Kitagawa Y, Ishihara R, Ishikawa H, Ito Y, Oyama T, Oyama T, Kato K, Kato H, Kawakubo H, Kawachi H, Kuribayashi S, Kono K, Kojima T, Takeuchi H, Tsushima T, Toh Y, Nemoto K, Booka E, Makino T, Matsuda S, Matsubara H, Mano M, Minashi K, Miyazaki T, Muto M, Yamaji T, Yamatsuji T, Yoshida M. Esophageal cancer practice guidelines 2022 edited by the Japan Esophageal Society: part 2. Esophagus. 2023 Jul;20(3):373-389. doi: 10.1007/s10388-023-00994-1. Epub 2023 Mar 30. No abstract available. PMID 36995449
- [Result] Li B, Chen H, Xiang J, Zhang Y, Kong Y, Garfield DH, Li H. Prevalence of lymph node metastases in superficial esophageal squamous cell carcinoma. J Thorac Cardiovasc Surg. 2013 Nov;146(5):1198-203. doi: 10.1016/j.jtcvs.2013.07.006. Epub 2013 Aug 26. PMID 23988285
- [Result] Ono S, Fujishiro M, Niimi K, Goto O, Kodashima S, Yamamichi N, Omata M. Long-term outcomes of endoscopic submucosal dissection for superficial esophageal squamous cell neoplasms. Gastrointest Endosc. 2009 Nov;70(5):860-6. doi: 10.1016/j.gie.2009.04.044. Epub 2009 Jul 4. PMID 19577748
- [Result] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593